CLINICAL TRIAL: NCT01885702
Title: Dendritic Cell Vaccination in Patients With Lynch Syndrome or Colorectal Cancer With MSI
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2008-005584-33
Record Dates: First submitted 2013-06-18; First posted 2013-06-25 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer
Keywords: Dendritic cell vaccination; MSI-high colorectal cancer (CRC); Vaccines; Immunotherapy; CRC; Germline MMR-gene mutation without disease criteria of CRC
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MSI-positive CRC patients (Experimental): I) Adjuvant DC vaccinations for MSI-positive CRC patients (n=5)
  Interventions: Biological: DC vaccination
- Carriers of germline MMR-gene mutation (Experimental): II) Preventive DC vaccinations for carriers of germline MMR-gene mutation (n=20) withhout manifestation of CRC
  Interventions: Biological: DC vaccination

INTERVENTIONS:
Biological: DC vaccination — DC vaccination

SUMMARY:
Objectives:

In this Radboud University Nijmegen Medical Centre (RUNMC) initiated study our first objective is to investigate toxicity (safety and feasibility) of vaccination with frameshift-derived neoantigen-loaded DC of CRC patients with an MSI-positive CRC and persons who are known to be carrier of a germline MMR-gene mutation with no signs of disease yet.

The secondary objectives of the study are:

* to demonstrate that peptide-loaded DC can induce or enhance an immune response to tumor-associated antigen CEA and specific frameshift-derived neoantigens in the study population.
* to study the pathological and clinical responses, e.g. disease-free survival, determined according to the standard protocol.

Study design:

This study is a phase I/II open-label study.

Study population:

Two groups of adults will be vaccinated:

Group I) CRC patients, who are known to carry a germline MMR-gene mutation and patients with an MSI-positive CRC and yet unknown or negative MMR-gene mutation status.

Group II) persons who are known to be carrier of a germline MMR-gene mutation with no signs of disease yet. All participants need to be HLA-A2.1 positive.

DETAILED DESCRIPTION:
Rationale of this study:

Ex vivo generated and tumor-antigen-loaded dendritic cells (DC) are currently used in clinical vaccination protocols in cancer patients. DC vaccines are safe, with minimal side effects. Evaluating more than 200 patients treated the past ten years we found that clinical responses measured in several patients directly coincide with specific cytotoxic T cell responses. The majority of studies investigated the therapeutic effects of DC vaccines in late-stage cancer patients with metastasis. In these (heavily) pretreated patients the immune system is compromised. Based on our observations that a specific immune response is indicative for a good clinical outcome we believe that the full potential of these immunostimulatory cells has to be exploited in high-risk patients with low tumor burden or in a precancerous state.

A good clinical model are carriers of a germline mutation in one of the DNA mismatch repair (MMR) genes, such as patients with Lynch syndrome (also known as Hereditary Non-Polyposis Colorectal Cancer or HNPCC). These persons have a lifetime risk of 60-80% for colorectal cancer that has developed within a few years from a precancerous adenoma. The immune system is thought to be of potential great importance as the colorectal cancer in Lynch syndrome is characterized by a strong lymphocyte infiltration, even at the stage of adenomas. In affected cancer lesions, MMR dysfunction results in frameshift mutations at short, repetitive DNA sequences referred to as microsatellites. In coding regions these mutations destroy gene function and have been demonstrated to lead to the production of neopeptides. These neopeptides are: 1) tumor specific, because frameshift mutations only occur in tumor cells and their premalignant progenitors, 2) are very similar between patients, since the same genes are affected by the mismatch repair defect and 3) immunogenic, since cytotoxic T cells (CTL) and helper T cells could be induced in vitro from blood of patients with Lynch syndrome. Similar mechanisms occur in sporadic colon cancer with MMR dysfunction, which represents about 10-15% of all colorectal 2.

Objectives:

In this Radboud University Nijmegen Medical Centre (RUNMC) initiated study our first objective is to investigate toxicity (safety and feasibility) of vaccination with frameshift-derived neoantigen-loaded DC of CRC patients with an MSI-positive CRC and persons who are known to be carrier of a germline MMR-gene mutation with no signs of disease yet.

The secondary objectives of the study are to demonstrate that peptide-loaded DC can induce or enhance an immune response to tumor-associated antigen CEA and specific frameshift-derived neoantigens in the study population. And we want to study the pathological and clinical responses, e.g. disease-free survival, determined according to the standard protocol.

Study design:

This study is a phase I/II open-label study.

Study population:

Two groups of adults will be vaccinated:

Group I) CRC patients, who are known to carry a germline MMR-gene mutation and patients with an MSI-positive CRC and yet unknown or negative MMR-gene mutation status.

Group II) persons who are known to be carrier of a germline MMR-gene mutation with no signs of disease yet. All participants need to be HLA-A2.1 positive.

Main study endpoints:

The first objective of this study is to toxicity (safety and feasibility) of vaccination with frameshift-derived neoantigen-loaded DC. This will be measured by recording of the adverse events according to the Common Terminology Criteria for Adverse Events version 3.0.

The secondary objectives of the study are to demonstrate that peptide-loaded DC can induce or enhance an immune response to tumor-associated antigen CEA and specific frameshift-derived neoantigens in the study population. Immune responses will be assessed as:

* proliferative and humoral response to KLH
* cytokine production of KLH stimulated PBMC
* tumor antigen-specific T cell responses in peripheral blood
* tumor antigen-specific T cell responses in biopsies from DTH
* cytokine production of T cells in biopsies from DTH
* cytotoxicity of T cells in biopsies from DTH
* immunohistochemical characterization of DTH infiltrating lymphocytes

The pathological and clinical responses, e.g. disease-free survival, will be determined according to the standard protocol.

ELIGIBILITY:
Inclusion Criteria:

* histologically documented evidence of CRC (group I) and Lynch syndrome carrier without signs of disease (group II)
* HLA-A2.1 phenotype is required
* MSI high tumor
* WBC >3.0 x 109/l, lymphocytes >0.8 x 109/l, platelets >100 x 109/l, serum crea¬tinine <150 µmol/l, serum bilirubin <25 µmol/l
* WHO performance status 0-1 (Karnofsky 100-70%)
* Age 18-75 years
* Expected adequacy of follow-up
* Written informed consent

Exclusion Criteria:

* History of malignancy in the past 5 years with the exception of adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix
* Serious active infections, HbsAg or HIV positive (test only in case of high risk or clinical suspicion)
* Autoimmune diseases or organ allografts
* Concomitant use of immunosuppressive drugs
* Known allergy to shell fish
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2010-10; Primary Completion 2016-04 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Safety and feasibility of vaccination with frameshift-derived neoantigen-loaded DC of CRC patients | 5 years
  Patients will be followed for toxicity, autoimmunity and immunological response during the study and 2 and 6 months thereafter at the outpatient clinic. Subsequently, follow up will be performed as for standard practice.
  Toxicity will be assessed using the Clinical Toxicity Criteria NCI CTC version 3.0.

SECONDARY OUTCOMES:
To evaluate whether peptide-loaded DC can induce or enhance an immune response to tumor-associated antigen CEA and specific frameshift-derived neoantigens in the study population | 5 years
Pathological responses | 5 years
  Pathological evaluation: Biopsies of carcinomas and or adenomas will be taken. One will be snap frozen and stored at -80 and one will be fixed in buffered formalin, for maximum of 24 hours and processed using microwave enhanced procedures. The composition of the tissue will be evaluated using standard histology supplemented with immunohistochemistry for subsets of inflammatory cells. The amount of and composition of the inflammation will be quantified using automated and semi automated quantitative methods. Based on initial results mRNA studies on cytokines and or chemokines will be performed and in addition immunohistochemistry for receptors for these molecules.
Clinical responses, e.g. disease-free survival, determined according to the standard protocol. | 5 years
  Progression-free survival is defined as the time from registration to the first recurrence of disease. Overall survival is defined as the time from registration to death. The status of disease is determined at regular intervals by taking the patients's history, physical examination, and colonoscopy. If signs or symptoms suggest disease recurrence at any site, the appropriate tests should be performed to confirm or exclude this.

CONTACTS AND LOCATIONS:
Overall Officials: Nicoline Hoogerbrugge-van der Linden, professor, Study Director — Radboud University Medical Center; Jolanda IM de Vries, professor, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared in an upcoming publication.